CLINICAL TRIAL: NCT03757481
Title: Long-term Outcome After Heparin and Edoxaban Versus Heparin Plus Vitamin K Antagonists for Acute Deep Vein Thrombosis and Pulmonary Embolism HOKUSAÏ POST VT
Brief Title: Long-term Outcome After Heparin and Edoxaban Versus Heparin Plus Vit K Antagonists for Acute DVT and PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL18_0005; UF 7548 (Other: Montpellier University Hospital)
Record Dates: First submitted 2018-11-23; First posted 2018-11-29 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Post Thrombotic Syndrome; Deep Vein Thrombosis; Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- no intervention (Other): patients with history of PE (pulmonary embolism) with acute DVT (deep veinous thrombosis) treated with heparin plus edoxaban or heparin plus warfarin
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — SF-36 questionnaire , PembQoL, Villalta score ,PembQoL

SUMMARY:
Centers that participated in the HOKUSAI VTE trial will be invited to collect follow of previously enrolled patients at least 2 years after the index VTE.

DETAILED DESCRIPTION:
HOKUSAI VTE trial was a randomised double blind non inferiority trial that compared the efficacy and safety of heparin ) (enoxaparin or unfractionated heparin) followed by edoxaban with heparin (enoxaparin or unfractionated heparin) followed by warfarin (target INR 2-3) in patients with acute, symptomatic VTE.

Centers that participated in the HOKUSAI VTE trial will be invited to collect follow of previously enrolled patients at least 2 years after the index VTE.

patients with index DVT will be asked to complete the SF-36 and PembQoL questionnaire to assess the (venous disease-specific) quality of life.

The Villalta score will be used to assess PTS. The objectively and subjectively obtained Villalta score- known as the patient reported Villalta -will be compared .

Among patients with with an index PE, the QoL will be assessed bu the validated generic (SF-36) and DVT at index will be examined for PTS and will be asked to complete all questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patient who participated in the HOKUSAI VTE trial

Exclusion Criteria:

* patient deprived of liberty
* patient under guardianship

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of PTS in patients with an acute DVT | 2 years
  PTS is defined by a Villalta index >5 or the presence of venous ulcer
PE related quality of life | 2 years after the index PE
  questionnaire SF 36

CONTACTS AND LOCATIONS:
Overall Officials: isabelle QUERE, PH, Principal Investigator — University Hospital, Montpellier
Locations (11):
- France (11):
  - Amiens University Hospital, Amiens
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Dijon University Hospital, Dijon
  - Grenoble University Hospital, Grenoble
  - Le Mans Hospital, Le Mans
  - Montpellier University Hospital, Montpellier
  - Nice University Hospital, Nice
  - APHP Hôpital Européen Georges Pompidou, Paris
  - Strasbourg University Hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bistervels IM, Bavalia R, Beyer-Westendorf J, Ten Cate-Hoek AJ, Schellong SM, Kovacs MJ, Falvo N, Meijer K, Stephan D, Boersma WG, Ten Wolde M, Couturaud F, Verhamme P, Brisot D, Kahn SR, Ghanima W, Montaclair K, Hugman A, Carroll P, Pernod G, Sanchez O, Ferrari E, Roy PM, Sevestre-Pietri MA, Birocchi S, Wik HS, Hutten BA, Coppens M, Naue C, Grosso MA, Shi M, Lin Y, Quere I, Middeldorp S; Hokusai PTS Investigators. Postthrombotic syndrome and quality of life after deep vein thrombosis in patients treated with edoxaban versus warfarin. Res Pract Thromb Haemost. 2022 Jul 1;6(5):e12748. doi: 10.1002/rth2.12748. eCollection 2022 Jul. PMID 35992565
- [Background] Bavalia R, Bistervels IM, Boersma WG, Quere I, Brisot D, Falvo N, Stephan D, Couturaud F, Schellong S, Beyer-Westendorf J, Montaclair K, Ghanima W, Ten Wolde M, Coppens M, Ferrari E, Sanchez O, Carroll P, Roy PM, Kahn SR, Meijer K, Birocchi S, Kovacs MJ, Hugman A, Ten Cate H, Wik H, Pernod G, Sevestre-Pietri MA, Grosso MA, Shi M, Lin Y, Hutten BA, Verhamme P, Middeldorp S; Hokusai post-PE study investigators. Quality of life in patients with pulmonary embolism treated with edoxaban versus warfarin. Res Pract Thromb Haemost. 2021 Jul 14;5(5):e12566. doi: 10.1002/rth2.12566. eCollection 2021 Jul. PMID 34278193